CLINICAL TRIAL: NCT00762892
Title: A Pilot Study--randomized, Prospective, Single Site Trial Evaluating Raltegravir vs. Atazanavir in Combination With Truvada® for the Treatment of Antiretroviral naïve HIV Infected Patients
Brief Title: Raltegravir vs. Atazanavir in Combination With Truvada® for the Treatment of Antiretroviral naïve HIV Infected Patients
Acronym: RAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tanvir K. Bell, MD, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: raltegravir atazanavir naive
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: HIV Infections
Keywords: Raltegravir; Integrase inhibitor; Protease inhibitor; Naive patients; HIV disease; Lipids; Treatment Naïve
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir (Active Comparator): Raltegravir in combination with truvada (tenofovir and emtricitabine)
  Interventions: Drug: Raltegravir and truvada
- Atazanavir (Active Comparator): Atazanavir, low dose ritonavir, and truvada (tenofovir and emtricitabine)
  Interventions: Drug: Atazanavir, Norvir and Truvada

INTERVENTIONS:
Drug: Raltegravir and truvada — Raltegravir 400 mg po bid, truvada 1 tab q daily
  Other Names: Truvada is tenofovir 300 mg and emtricitabine 200 mg
  Arms: Raltegravir
Drug: Atazanavir, Norvir and Truvada — Atazanavir 300 mg po q daily, Norvir 100 mg po q daily and Truvada 1 tablet po q daily
  Other Names: Truvada is tenofovir 300 mg and emtricitabine 200 mg
  Arms: Atazanavir

SUMMARY:
This is a pilot that will evaluate two regimens for treating HIV infected patients that haven't been on treatment before. HIV/AIDS patients may have an increased risk of myocardial infarction and antiretroviral therapy used may contribute to this. We will evaluate virological, immunological and cardiovascular effects of two HIV treatment regimens.

DETAILED DESCRIPTION:
We will check blood studies used to evaluate HIV patients response to therapy including CD4 count and HIV viral load test. We will check routine safety labs done on HIV patients and also check homocysteine levels and creatine kinase level. We will evaluate homocysteine and IL6 levels at baseline, week 48, and week 96.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be HIV-1 positive and naïve to HIV therapy.
* Patients must plan to participate and be available for the trial for the 96-week study period.
* Patients followed at Thomas Street Clinic.
* Patients must be over 18 years old.

Exclusion Criteria:

* Patients must not be pregnant or plan to become pregnant over the 96-week study period.
* Patients cannot be on a proton pump inhibitor.
* Patients cannot be undergoing treatment for active tuberculosis.
* Renal Insufficiency with a creatinine clearance < 50 ml/min/1.73 m2 by the MDRD GFR calculation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanvir K Bell, MD, Principal Investigator — UT-Houston
Locations (1):
- Thomas Street Clinic, Houston, Texas, United States

REFERENCES:
- See also: open access journal — http://omicsonline.org/lipid-and-biomarker-differences-between-raltegravir-and-atazanavir-ritonavir-at-48-weeks-in-the-raltegravir-atazanavir-2155-6113.1000192.php?aid=11665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: approached patients HIV positive, naive to therapy, single site, English and Spanish speaking/writing.
Period: Overall Study
Arm/Group | Raltegravir | Atazanavir
Started | 14 | 14
Completed | 9 | 8
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Incarceration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir | Atazanavir | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 40.7 (11) | 38.8 (10) | 39.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in CD4 Count at 48 Weeks
Time Frame: Baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Raltegravir | Atazanavir
Number analyzed (Participants) | 9 | 8
cells/uL | 192 (26) | 205 (27)

2. Secondary Outcome: Change From Baseline in Lipids at 48 Weeks
Time Frame: Baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Raltegravir | Atazanavir
Number analyzed (Participants) | 9 | 8
mg/dL
  Total cholesterol | -0.25 (7.66) | 8.13 (11.96)
  Triglycerides | -15.50 (18.47) | 16.88 (40.89)
  HDL cholesterol | -1.5 (2.58) | -1.38 (3.08)
  LDL cholesterol | 4.13 (7.54) | 5.88 (14.46)

3. Primary Outcome: Change From Baseline in Log HIV Viral Load at 48 Weeks
Time Frame: Baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Raltegravir | Atazanavir
Number analyzed (Participants) | 9 | 8
copies/mL | -3.05 (0.28) | -3.29 (0.26)

4. Secondary Outcome: Change From Baseline in Interleukin-6 (IL-6) at 48 Weeks
Time Frame: Baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Raltegravir | Atazanavir
Number analyzed (Participants) | 9 | 8
pg/mL | -2.71 (1.63) | -4.47 (2.51)

5. Secondary Outcome: Change From Baseline in Homocysteine at 6 Months
Time Frame: Baseline and 48 weeks
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Raltegravir | Atazanavir
Number analyzed (Participants) | 9 | 8
umol/L | 0.53 (0.83) | 0.10 (0.94)

ADVERSE EVENTS:
Arm/Group | Raltegravir | Atazanavir
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=14) | Atazanavir (N=14)
MAI infection, multi-organ failure, death (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations are the relatively small sample size and loss to follow-up. Medical records of patients that were lost to follow up was reviewed to ensure that no SAE occurred. We also attempted multiple times to contact patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No